CLINICAL TRIAL: NCT00893880
Title: A Dose Response Trial to Evaluate Clinical and Mycological Effect of Nitric Oxide in Subjects With Tinea Pedis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nitric BioTherapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP8
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Last update posted 2012-10-22 (Estimated); Status verified 2012-10

CONDITIONS: Tinea Pedis
Keywords: Tinea Pedis; Athletes Foot; Nitric Oxide
MeSH Terms: conditions — Tinea Pedis | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): (1) 30min treatment
  Interventions: Drug: 1% gaseous Nitric Oxide blended in Oxygen
- 2 (Experimental): (1) 60min treatment
  Interventions: Drug: 1% gaseous Nitric Oxide blended in Oxygen
- 3 (Experimental): (2) 30min treatments over two consecutive days.
  Interventions: Drug: 1% gaseous Nitric Oxide blended in Oxygen
- 4 (Experimental): (2) 60min treatments over two consecutive days.
  Interventions: Drug: 1% gaseous Nitric Oxide blended in Oxygen

INTERVENTIONS:
Drug: 1% gaseous Nitric Oxide blended in Oxygen — 1% gaseous nitric oxide blended in oxygen applied for 30-60 minutes over 1-2 consecutive days.

SUMMARY:
A multi-arm trial to evaluate the efficacy and safety of using gaseous nitric oxide to treat moderate to severe tinea pedis.

ELIGIBILITY:
Inclusion Criteria:

* Positive clinical findings (moderate to severe, indicated by a CSSS ≥ 6) for interdigital or bullous tinea pedis as determined by clinical examination (subjects with moccasin symptoms in addition to above may also be included at the discretion of the investigator).
* Written informed consent must be obtained from the subject.
* Must ≥ 18 years of age, unless local laws dictate otherwise.
* Must agree to avoid professional pedicures or application of any nail polish product or nail cosmetic to the toenails after the screening visit until the conclusion of the trial.
* Must not be pregnant or nursing, and if of childbearing potential, agree to take measures to avoid pregnancy during the study period

Exclusion Criteria:

* Has a diagnosis of either psoriasis or eczema, in or immediately around the area under evaluation.
* Has a visual diagnosis, by the investigator, of onychomycosis at a level, which in the opinion of the investigator would compromise the integrity of the study.
* Use of topical antifungals e.g. (clotrimazole, ketoconazole,miconazole, oxiconazole- (Oxistat®, Glaxo Smith Kline), sulconazole, naftifine (Naftin®, Merz), terconazole, econazole nitrate (Spectazole®, Ortho-McNeil), butoconazole ,Fluconazole, ciclopirox olamine-(Loprox®, Medicis), tolnaftate, haloprogin), Zeasorb-AF , antibacterials and corticosteroids in the preceding 14 days of screening visit (Day 1), on or immediately around the area under evaluation.
* Use of oral or injectable systemic corticosteroids in the preceding 7 or 30 days respectively, of screening visit (Day 1)
* Use of systemic antifungals in the preceding 30 days of screening visit (Day1) including - (terbinafine - (Lamisil®, Novartis), Itraconazole - (Sporanox®, Janssen), fluconazole- (Diflucan®, Pfizer), ketoconazole, miconazole, griseofulvin (Gris-PEG®, Pedinol), butoconazole, terconazole, Potassium iodide)
* Has used any investigational drug(s) within 30 days preceding screening visit (Day 1)
* Is pregnant or is a nursing mother
* Is a woman of child bearing potential who is not using an adequate form of contraception (or abstinence)
* Is < 18 years of age, unless local laws dictate otherwise.
* Is immunosuppressed (undergoing chemotherapy, neutropenia (PMNs , < 500/mm3), HIV with CD4+ < 200/mm3.
* Suffers from a condition, which, in the opinion of the medical investigator, would compromise his/her safety and / or the quality of the data. Such conditions may include collagen vascular disease, diabetes mellitus, Cushing's Disease, hematological malignancy, chronic mucocutaneous candidiasis or atopy STATISTICS This clinical evaluation is intended to demonstrate

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2009-06; Primary Completion 2010-01 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Complete cure (negative KOH and culture and no signs or symptoms), Effective treatment (negative KOH and culture and at most mild erythema or scaling), Negative mycology (negative KOH and culture). | 29 days

SECONDARY OUTCOMES:
Determine the clinical and mycological effect of 1% gaseous nitric oxide (gNO) as a treatment for Tinea Pedis in the clinically evaluable population at the Test-of-Cure (TOC) evaluation (4 weeks post-treatment) according to the definitions below: | 29 days
Determine the clinical and mycological effect of the topical application of 1% gNO as confirmed by pre treatment positive culture and clinical signs and symptoms compared to 2 weeks post treatment outcomes according to definitions below: | 14 days
Determine the clinical and mycological effect of the topical application of 1% gNO as confirmed by pre treatment positive culture and clinical signs and symptoms compared to 1 week post treatment outcomes according to definitions below: | 7 days
Determine the safety of daily topical applications of 1% gNO as confirmed by methemoglobin levels and adverse events. | 29 days

CONTACTS AND LOCATIONS:
Locations (4):
- Mediprobe Research, Inc, London, Ontario, Canada
- Saint Kitts and Nevis (3):
  - Eureka Health Services, Ramsbury Site, Nevis
  - Diversified Healthcare Solutions, Basseterre, Saint Kitts
  - Medical Associates, Basseterre, Saint Kitts